CLINICAL TRIAL: NCT03662074
Title: Phase II Pilot Study of Subsequent Line Gemcitabine and Nivolumab for Advanced SCLC
Brief Title: Subsequent Line Gemcitabine and Nivolumab in Treating Participants With Metastatic Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After interim analysis decided not to move forward with continuing the trial.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00051024; NCI-2018-01803 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 62418 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Results first posted 2021-11-12 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Small Cell Lung Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Gemcitabine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (gemcitabine, nivolumab) (Experimental): Participants receive gemcitabine IV over 30 minutes and nivolumab IV over 60 minutes on day 1. Treatment repeats every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Gemcitabine; Biological: Nivolumab

INTERVENTIONS:
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II pilot trial studies how well gemcitabine and nivolumab work in treating participants with small cell lung cancer that has spread to other parts of the body after other treatments have failed. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. Giving second-line gemcitabine and nivolumab may work better in treating participants with small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare response rate (RR) of gemcitabine and nivolumab (G+N) after 4 cycles (8 weeks) to historical controls treated with nivolumab alone.

SECONDARY OBJECTIVES:

I. To compare median overall survival (OS) of G+N to historical controls treated with nivolumab alone.

II. To compare median progression-free survival (PFS) of G+N to historical controls treated with nivolumab alone.

III. To evaluate for tolerability of G+N at each treatment cycle and then every 8 weeks after treatment is completed.

EXPLORATORY OBJECTIVES:

I. To correlate immunophenotypic changes among lymphocytes (quantitative measurements of CD4 and CD8 T-cells) with radiographic response and overall survival before treatment, after treatment and between 8-12 weeks after treatment.

II. Among those patients with tumor mutation burden (TMB) status available, to describe the association between TMB (low, medium, or high) and RR, OS, and PFS.

III. Assess the patient perspective of symptomatic adverse events using self-reported items from the National Cancer Institute (NCI) Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE).

OUTLINE:

Participants receive gemcitabine intravenously (IV) over 30 minutes and nivolumab IV over 60 minutes on day 1. Treatment repeats every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days, 6-10 weeks, and every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed incurable SCLC and have had prior treatment with platinum-based chemotherapy. High-grade neuroendocrine tumors that are suspected to be of bronchopulmonary origin can be enrolled if they have had prior treatment with a SCLC chemotherapy regimen (e.g. platinum plus etoposide).
* Patients should not be demonstrating end-organ damage due to rapid progression of disease based on the most recent assessment of the treating physician.
* Patients must have radiographically measurable metastatic disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Absolute neutrophil count >= 1,500/mcL.
* Platelets >= 100,000/mcL.
* Chemotherapy agents are known to be teratogenic, therefore women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document.

Exclusion Criteria:

* Patients who have previously received either gemcitabine or an immune checkpoint inhibitor can be enrolled.
* Emergent need for palliative radiation.
* Patients may not be receiving any other investigational agents for the treatment of nonsmall cell lung cancer.
* History of allergic reaction to gemcitabine.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects with chemotherapy. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy, breastfeeding should be discontinued.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W. Lycan, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Gemcitabine, Nivolumab)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Gemcitabine, Nivolumab)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Responses to Therapy Per Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Objective RR (complete response [CR] + partial response [PR]) will be compared between this study sample and a historical benchmark value of 10%. For this comparison we will use a one-sample test of proportion.
  * Complete Response (CR): Disappearance of all target lesions.
  * Partial Response (PR): Decrease by ≥ 30% in sum of longest diameter of target lesions.
  * Stable Disease (SD): Not meeting criteria for CR, PR, or PD.
  * Progressive Disease (PD): Increase by ≥ 20% in sum of longest diameter of target lesions or the appearance of one or more new lesions.
  The response in non-target lesions is defined as follows:
  * Complete Response (CR): Complete disappearance of all non-target lesions.
  * Stable Disease (SD): Persistence of one or more non-target lesion(s).
  * Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Gemcitabine, Nivolumab)
Number analyzed (Participants) | 14
Participants
  Partial response | 1
  Progressive disease | 11
  Lost to follow up | 2
Statistical Analysis 1: Comparison: Treatment (Gemcitabine, Nivolumab); Test type: Other; The pre-specified analysis plan as per the protocol is to proceed to the second stage of recruitment for additional participants if the response proportion exceeds the historical control of 10%

2. Secondary Outcome: Overall Survival (OS) - Number of Participants
Description: OS will be estimated using standard Kaplan Meier survival analysis methods.
Time Frame: Duration of time from the start of treatment to date of death, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Gemcitabine, Nivolumab)
Number analyzed (Participants) | 14
Participants
  Deaths - any reason | 8
  Survivors | 6

3. Secondary Outcome: Overall Survival (OS) - Months
Description: A median value (months) of overall survival will be estimated using standard Kaplan Meier survival analysis methods.
Time Frame: Duration of time from the start of treatment to date of death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Gemcitabine, Nivolumab)
Number analyzed (Participants) | 14
months | 3.2 [1.7 to 9.2]

4. Secondary Outcome: Progression-free Survival (PFS) - Number of Participants
Description: Progression-free survival will be estimated using standard Kaplan Meier survival analysis methods. Progression-Free Survival (PFS) is defined as the duration of time from the start of treatment to the time of investigator assessed progression or death. Progressive Disease (PD): Increase by ≥ 20% in sum of longest diameter of target lesions or the appearance of one or more new lesions
Time Frame: Duration of time from the start of treatment to the time of investigator assessed progression or death, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Gemcitabine, Nivolumab)
Number analyzed (Participants) | 14
Participants
  Participants that had disease progression | 11
  Participants that did not have disease progression | 3

5. Secondary Outcome: Progression-free Survival (PFS) - Months
Description: A median value (months) of progressive-free survival will be estimated using standard Kaplan Meier survival analysis methods. Progressive Disease (PD): Increase by ≥ 20% in sum of longest diameter of target lesions or the appearance of one or more new lesions
Time Frame: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Gemcitabine, Nivolumab)
Number analyzed (Participants) | 14
months | 1.8 [1.6 to 8.6]

6. Secondary Outcome: Number of Adverse Events
Description: Toxicity rates will be estimated by responder status and presented overall and by body site per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time Frame: Up to 2 years
Measure: Number; unit: Number of adverse events reported
Arm/Group | Treatment (Gemcitabine, Nivolumab)
Number analyzed (Participants) | 14
Number of adverse events reported | 12

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment (Gemcitabine, Nivolumab)
All-Cause Mortality (participants affected / at risk) | 8/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Gemcitabine, Nivolumab) (N=14)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Gemcitabine, Nivolumab) (N=14)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT03662074/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT03662074/ICF_001.pdf